CLINICAL TRIAL: NCT04271644
Title: BCMA-Targeted CAR-T Cell Therapy for Relapsed/Refractory Multiple Myeloma and Plasma Cell Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC002
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma; Neoplasm, Plasma Cell; Multiple Myeloma in Relapse
Keywords: Multiple Myeloma; BCMA; Chimeric Antigen Receptor T Cell
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCMA CAR-T cells treat (Experimental): Patients will be be treated with BCMA CAR-T cells
  Interventions: Biological: BCMA CAR-T cells

INTERVENTIONS:
Biological: BCMA CAR-T cells — BCMA CAR-T cell therapy

SUMMARY:
This is a single arm study to evaluate the efficacy and safety of BCMA-targeted CAR-T cells therapy for patients with relapsed/refractory Multiple Myeloma.

DETAILED DESCRIPTION:
There are limited options for treatment of relapse/refractory Multiple Myeloma. BCMA is expressed on most Multiple Myeloma cells so it is an ideal target for CAR-T. In this study, investigators will evaluate the safety and efficacy of CAR-T targeting BCMA in patients with relapsed/refractory Multiple Myeloma. The primary goal is safety and efficiency assessment, including adverse events and disease status after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent;
2. Diagnose as relapsed /refractory multiple myeloma or other plasma cell disease, and meet one of the following conditions:

   1. Failed to standard chemotherapy regimens;
   2. Relapse after complete remission, high-risk and / or refractory patients ;
   3. Relapse after hematopoietic stem cell transplantation;
3. Evidence for cell membrane BCMA expression；
4. All genders, ages: 18 to 75 years；
5. The expect time of survive is above 3 months;
6. KPS>60；
7. No serious mental disorders ;
8. Left ventricular ejection fraction ≥50%
9. Sufficient hepatic function defined by ALT/AST≤3 x ULN and bilirubin≤2 x ULN;
10. Sufficient renal function defined by creatinine clearance≤2 x ULN;
11. Sufficient pulmonary function defined by indoor oxygen saturation≥92%;
12. With single or venous blood collection standards, and no other cell collection contraindications;
13. Ability and willingness to adhere to the study visit schedule and all protocol requirements.

Exclusion Criteria:

1. Previous history of other malignancy;
2. Presence of uncontrolled active infection;
3. Evidence of disorder that need the treatment by glucocorticoids;
4. Active or chronic GVHD；
5. The patients treatment by inhibitor of T cell；
6. Pregnant or breasting-feeding women;
7. Any situation that investigators regard not suitable for attending in this study (e.g. HIV , HCVinfection or intravenous drug addiction) or may affect the data analysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events that related to treatment | 2 years
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
The response rate of BCMA CAR-T treatment in patients with relapse/refractory Multiple Myeloma that treatment by BCMA CAR-T cells therapy | 2 years
  The response rate of BCMA CAR-T treatment will be recorded and assessed according to the IMWG

SECONDARY OUTCOMES:
Rate of BCMA CAR-T cells in bone marrow and peripheral blood | 2 years
  In vivo (bone marrow and peripheral blood) rate of BCMA CAR-T cells were determined by means of flow cytometry
Quantity of BCMA CAR copies in bone marrow and peripheral blood | 2 years
  In vivo (bone marrow and peripheral blood) quantity of BCMA CAR copies were determined by means of qPCR
Quantity of clonal plasma cells in bone marrow | 1 years
  In vivo (bone marrow) quantity of clonal plasma cells
Levels of Cytokines in Serum | 1 years
  In vivo (Serum) quantity of cytokines
Duration of Response (DOR) of BCMA CAR-T treatment in patients with refractory/relapsed multiple myeloma | 2 years
  DOR will be assessed from the first assessment of sCR/CR/VGPR/PR to the first assessment of recurrence or progression of the disease or death from any cause (censored)
Progress-free survival(PFS) of BCMA CAR-T treatment in patients with refractory/relapsed multiple myeloma | 2 years
  PFS will be assessed from the first CAR-T cell infusion to death from any cause or the first assessment of progression (censored)
Overall survival(OS) of BCMA CAR-T treatment in patients with refractory/relapsed multiple myeloma | 2 years
  OS will be assessed from the first CAR-T cell infusion to death from any cause (censored)

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, MD, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China; Cheng Qian, PhD, Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- 920th Hospital of Joint Logistics Support Force, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No